CLINICAL TRIAL: NCT01006616
Title: A 2-Year, Dose Range-Finding, Adaptive-Design Study of the Effects of SCH 527123 in Subjects With Moderate to Severe COPD
Brief Title: Long-Term Study of the Effects of Navarixin (SCH 527123, MK-7123) in Participants With Moderate to Severe COPD (MK-7123-019)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05575; 2008-003780-38 (EudraCT Number); P05575 (Other: Merck Research Laboratories)
Record Dates: First submitted 2009-10-01; First posted 2009-11-03 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — navarixin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Navarixin 10 mg (Experimental): Participants receive navarixin 10 mg, as one navarixin 10 mg capsule and two placebo capsules, administered orally once daily (QD) for up to 2 years
  Interventions: Drug: Navarixin; Drug: Placebo; Drug: Rescue medication
- Navarixin 30 mg (Experimental): Participants receive navarixin 30 mg, as one navarixin 30 mg capsule and two placebo capsules, administered orally QD for up to 2 years
  Interventions: Drug: Navarixin; Drug: Placebo; Drug: Rescue medication
- Navarixin 50 mg (Experimental): Participants receive navarixin 50 mg, as two navarixin 10 mg capsules and one navarixin 30 mg capsule, administered orally QD for up to 2 years
  Interventions: Drug: Navarixin; Drug: Rescue medication
- Placebo (Placebo Comparator): Participants receive placebo to navarixin, as three placebo capsules, administered orally QD for up to 2 years
  Interventions: Drug: Placebo; Drug: Rescue medication

INTERVENTIONS:
Drug: Navarixin — Navarixin 10 mg and 30 mg capsules
  Arms: Navarixin 10 mg; Navarixin 30 mg; Navarixin 50 mg
Drug: Placebo — Placebo to navarixin capsules
  Arms: Navarixin 10 mg; Navarixin 30 mg; Placebo
Drug: Rescue medication — Short-acting β-agonist (SABA), anticholinergic, or a combination SABA/anticholinergic

SUMMARY:
Neutrophils are thought to play an important role in the pathophysiology of chronic obstructive pulmonary disease (COPD). Navarixin (SCH 527123, MK-7123) is an antagonist of the cysteine-X-cysteine chemokine receptor 2 (CXCR2) and is thought to reduce neutrophil migration to the diseased lung. It is theorized that reducing neutrophil migration to the diseased lung will improve a participant's symptoms and the natural history of the disease.

The study will consist of a 2-week screening period followed by a 2-year (104-week) double-blind treatment period. The 2-year Treatment Period will be made up of two phases: a 26-week (6-month) dose range-finding phase with 3 active arms and 1 placebo arm (Period 1), followed by a 78-week (18-month) long-term safety and efficacy phase (Period 2). Participants participating in the original 6-month study (Period 1) may elect not to continue into the 18-month extension study (Period 2).

Hypothesis: navarixin, 50 mg, or the highest remaining dose if the 50-mg dose is discontinued, is superior to placebo with respect to improving airflow.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD for at least 2 years based on American Thoracic Society/European Respiratory Society (ATS/ERS) current guidelines or symptoms consistent with COPD for at least 2 years.
* >40 to <=75 years of age, of either sex, and of any race.
* No exacerbation or respiratory infection in the past 6 weeks.
* Smoker or ex-smoker with more than 10 pack-year history.

Exclusion Criteria:

* Diagnosis of asthma or other clinically relevant lung disease (other than COPD), i.e., sarcoidosis, tuberculosis, pulmonary fibrosis, severe bronchiectasis, or lung cancer.
* Significant X-ray findings.
* Use of supplemental oxygen for >12 hours/day.

Ages: 41 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2011-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Rennard SI, Dale DC, Donohue JF, Kanniess F, Magnussen H, Sutherland ER, Watz H, Lu S, Stryszak P, Rosenberg E, Staudinger H. CXCR2 Antagonist MK-7123. A Phase 2 Proof-of-Concept Trial for Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2015 May 1;191(9):1001-11. doi: 10.1164/rccm.201405-0992OC. PMID 25695403
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P05575&kw=7123-019&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Period 1 (6 Months)
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Started | 152 | 156 | 153 | 155
Treated | 152 | 156 | 152 | 154
Completed | 126 | 102 | 102 | 128
Not Completed | 26 | 54 | 51 | 27
Not completed — Adverse Event | 10 | 31 | 37 | 9
Not completed — Lack of Efficacy | 3 | 4 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrew, Reason Unrelated to Treatment | 6 | 5 | 2 | 3
Not completed — Withdrew, Reason Related to Treatment | 0 | 3 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 2 | 2 | 0
Not completed — Did Not Meet Protocol Eligibility | 5 | 7 | 5 | 5
Not completed — Noncompliance With Protocol | 0 | 2 | 2 | 3
Not completed — Not Treated | 0 | 0 | 1 | 1
Period: Period 2 (18 Months)
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Started | 75 (Period 2 was optional. Not all participants completing Period 1 continued into Period 2.) | 63 (Period 2 was optional. Not all participants completing Period 1 continued into Period 2.) | 55 (Period 2 was optional. Not all participants completing Period 1 continued into Period 2.) | 82 (Period 2 was optional. Not all participants completing Period 1 continued into Period 2.)
Treated | 75 | 63 | 55 | 82
Completed | 0 | 0 | 0 | 0
Not Completed | 75 | 63 | 55 | 82
Not completed — Adverse Event | 6 | 6 | 6 | 4
Not completed — Lack of Efficacy | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Withdrew, Reason Unrelated to Treatment | 3 | 0 | 3 | 2
Not completed — Withdrew, Reason Related to Treatment | 0 | 6 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 4 | 0 | 1
Not completed — Noncompliance With Protocol | 0 | 1 | 0 | 1
Not completed — Study Terminated | 63 | 46 | 44 | 70

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population consists of all treated participants (1 participant in the Navarixin 50 mg group and 1 participant in the Placebo group did not receive study drug).
Groups:
- Navarixin 10 mg: Participants receive navarixin 10 mg, as one navarixin 10 mg capsule and two placebo capsules, administered orally QD for up to 2 years
- Total: Total of all reporting groups
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo | Total
Number analyzed (Participants) | 152 | 156 | 152 | 154 | 614
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.7 (6.9) | 63.2 (7.4) | 61.3 (7.5) | 63.3 (7.2) | 62.9 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 52 | 50 | 46 | 176
  Male | 124 | 104 | 102 | 108 | 438

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Post-bronchodilator Forced Expiratory Volume in 1 Second (FEV1) (Period 1)
Description: FEV1, as measured in liters by spirometry, is the amount of air expired in 1 second. Participants were assessed for post-bronchodilator FEV1 30 minutes after bronchodilator administration (4 puffs of albuterol/salbutamol or equivalent separated by 30-second intervals) (reversibility test) at Baseline and Week 26.
Time Frame: Baseline and Week 26
Population: The Full Analysis Set (FAS) population consisted of all participants who received at least one dose of study drug and had a Baseline and Week 26 assessment for post-bronchodilator FEV1.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 124 | 105 | 102 | 127
Liters | -0.009 (0.022) | -0.068 (0.023) | 0.028 (0.024) | -0.039 (0.022)
Statistical Analysis 1: Comparison: Navarixin 10 mg vs Placebo; Test type: Superiority or Other; p = 0.325, Constrained Longitudinal Data Analysis; Model with treatment, time, treatment by time interaction, and baseline smoking status (yes/no) and inhaled corticosteroid (ICS) use (yes/no); Mean Difference (Net) = 0.031, 95% CI 2-sided [-0.030 to 0.091]
Statistical Analysis 2: Comparison: Navarixin 30 mg vs Placebo; Test type: Superiority or Other; p = 0.370, Constrained Longitudinal Data Analysis; Model with treatment, time, treatment by time interaction, and baseline smoking status (yes/no) and ICS use (yes/no); Mean Difference (Net) = -0.029, 95% CI 2-sided [-0.091 to 0.034]
Statistical Analysis 3: Comparison: Navarixin 50 mg vs Placebo; Test type: Superiority or Other; p = 0.037, Constrained Longitudinal Data Analysis; Model with treatment, time, treatment by time interaction, and baseline smoking status (yes/no) and ICS use (yes/no); Mean Difference (Net) = 0.067, 95% CI 2-sided [0.004 to 0.131]

2. Primary Outcome: Percentage of Participants With an Adverse Event (AE) Related to a Blood Absolute Neutrophil Count (ANC) of Less Than 1.5x10^9 Cells/L
Description: The percentage of participants who experienced an AE related to an ANC of less than 1.5x10^9 cells/L at one or more visits during the first 26 weeks, the first 52 weeks and the first 104 weeks was to be calculated.
Time Frame: Up to 104 weeks
Population: The All Subjects as Treated (ASaT) population consisted of all participants who received at least one dose of study drug. The study was terminated during Period 2; no data were analyzed for this endpoint for up to 52 and up to 104 weeks.
Measure: Number; unit: Percentage of Participants
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 152 | 156 | 152 | 154
Percentage of Participants
  Up to Week 26 (n=152, 156, 152,154) | 3.3 | 12.8 | 20.4 | 0.6
  Up to Week 52 (n=0, 0, 0, 0) | NA — Study terminated; data not collected. | NA — Study terminated; data not collected. | NA — Study terminated; data not collected. | NA — Study terminated; data not collected.
  Up to Week 104 (n=0, 0, 0, 0) | NA — Study terminated; data not collected. | NA — Study terminated; data not collected. | NA — Study terminated; data not collected. | NA — Study terminated; data not collected.
Statistical Analysis 1: Comparison: Navarixin 10 mg vs Placebo; Test type: Superiority or Other; p = 0.096, Miettinen and Nurminen; Difference in percentages = 2.6, 95% CI 2-sided [-0.6 to 6.9] — Analysis of Week 26 data
Statistical Analysis 2: Comparison: Navarixin 30 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen; Difference in percentages = 12.2, 95% CI 2-sided [7.4 to 18.4] — Analysis of Week 26 data
Statistical Analysis 3: Comparison: Navarixin 50 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen; Difference in percentages = 19.7, 95% CI 2-sided [13.8 to 26.9] — Analysis of Week 26 data

3. Secondary Outcome: Change From Baseline in Post-bronchodilator FEV1 (Period 2)
Description: FEV1, as measured in liters by spirometry, is the amount of air expired in 1 second. Participants were to be assessed for post-bronchodilator FEV1 30 minutes after bronchodilator administration (4 puffs of albuterol/salbutamol or equivalent separated by 30-second intervals) (reversibility test) at Baseline, Week 52 and Week 104.
Time Frame: Baseline and Week 52, Week 104
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Baseline and Week 52 or Week 104 assessment for post-bronchodilator FEV1 in Period 2. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 66 | 47 | 44 | 65
Liters
  Week 52 (n=66, 47, 44, 65) | -0.047 (0.027) | -0.084 (0.031) | 0.028 (0.032) | -0.031 (0.027)
  Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

4. Secondary Outcome: Number of Participants With a Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: COPD exacerbation is defined as any deterioration of symptoms that leads to an increase in bronchodilator use on 2 or more consecutive days, or administration (at investigator's discretion) of antibiotics and/or systemic corticosteroids (above participant's usual dose), or an unscheduled COPD-related doctor visit, hospitalization or emergency room treatment. The numbers of participants who experienced at least one moderate to severe COPD exacerbation during the first 26 weeks, the first 52 weeks and the first 104 weeks of treatment were to be summarized.
Time Frame: Up to 26 , 52 and 104 weeks
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Week 26, Week 52 or Week 104 assessment for COPD exacerbation. The study was terminated during Period 2; no data were collected for this endpoint for up to 104 weeks.
Measure: Number; unit: Participants
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 152 | 156 | 152 | 154
Participants
  Up to Week 26 (n=152, 156, 152, 154) | 40 | 50 | 45 | 48
  Up to Week 52 (n=152, 156, 152, 154) | 50 | 58 | 51 | 53
  Up to Week 104 (n=0, 0, 0, 0) | NA — Study terminated; data not collected. | NA — Study terminated; data not collected. | NA — Study terminated; data not collected. | NA — Study terminated; data not collected.

5. Secondary Outcome: Percentage of Participants With a Moderate to Severe COPD Exacerbation
Description: COPD exacerbation is defined as any deterioration of symptoms that leads to an increase in bronchodilator use on 2 or more consecutive days, or administration (at investigator's discretion) of antibiotics and/or systemic corticosteroids (above participant's usual dose), or an unscheduled COPD-related doctor visit, hospitalization or emergency room treatment. The percentages of participants who experienced at least one moderate to severe COPD exacerbation during the first 26 weeks, the first 52 weeks and the first 104 weeks of treatment were to be summarized.
Time Frame: Up to 26, 52 and 104 weeks
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Baseline and Week 26, Week 52 or Week 104 assessment for COPD exacerbation. The study was terminated during Period 2; no data were collected for this endpoint for up to 104 weeks.
Measure: Number; unit: Percentage of Participants
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 152 | 156 | 152 | 154
Percentage of Participants
  Up to Week 26 (n=152, 156, 152, 154) | 26.3 | 32.1 | 29.6 | 31.2
  Up to Week 52 (n=152, 156, 152, 154) | 32.9 | 37.2 | 33.6 | 34.4
  Up to Week 104 (n=0, 0, 0, 0) | NA — Study terminated; data not collected. | NA — Study terminated; data not collected. | NA — Study terminated; data not collected. | NA — Study terminated; data not collected.

6. Secondary Outcome: Total Exacerbations of Chronic Pulmonary Disease Tool-Patient-Recorded Outcome (EXACT-PRO) Questionnaire Score
Description: The total score on the EXACT-PRO questionnaire is used to determine the frequency, severity, and duration of exacerbations of COPD. The 14-item EXACT-PRO questionnaire was to be completed by participants every evening to describe their experience of COPD during that day. Assessments were included for Breathlessness (5 items), Cough and Sputum (2 items), Chest Symptoms (3 items), and 4 additional items (Difficulty with Sputum, Tired or Weak, Sleep Disturbance, and Psychological State). Each item was measured on a 5- or 6-point scale. The total EXACT-PRO questionnaire score could range from 0 to 100, with a higher score indicating a more severe health state.
Time Frame: At 26, 52 and 104 weeks
Population: The FAS population was to consist of all participants who received at least one dose of study drug and had a Baseline and Week 26, Week 52 or Week 104 assessment for total EXACT-PRO score. This analysis was not conducted if results for percentage of participants with moderate to severe COPD exacerbation suggested no need for further investigation.
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Induced Sputum Absolute Neutrophil Counts
Description: Induced sputum samples were to be obtained from participants via the nebulized method for analysis of absolute neutrophil counts at Week 26, Week 52 and Week 104. The reported Baseline least squares (LS) means and standard deviations (SDs) are pooled across all treatment groups. The rationale for the use of pooled Baseline LS mean and SD values is the assumption that the Baseline LS mean and SD values are similar across treatment groups. The reported post-Baseline SDs are pooled across all treatment groups. The rationale for the use of an analysis of variance (ANOVA) method using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline, Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants at selected sites who received at least one dose of study drug and had a baseline and Week 26, Week 52 or Week 104 assessment for sputum neutrophil count. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 30 | 29 | 33 | 33
10^9 cells/L
  Baseline (n=30, 29, 33, 33) | 1.485 (0.706) | 1.485 (0.706) | 1.485 (0.706) | 1.485 (0.706)
  Week 26 (n=23, 13, 13, 17) | 1.763 (0.736) | 2.073 (0.736) | 0.860 (0.736) | 2.121 (0.736)
  Week 52 (n=9, 8, 3, 3) | 2.884 (0.462) | 2.022 (0.462) | 1.253 (0.462) | 3.218 (0.462)
  Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

8. Secondary Outcome: Change From Baseline in St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C) Total Score
Description: The SGRQ-C consists of 40 items aggregated into 3 component scores: Symptoms (frequency/severity), Activity (limited by breathlessness), Impacts (social functioning, psychological disturbances), and a Total score. Each response to a question is assigned a weight. Component scores are calculated by summing the weights from all positive items in that component, dividing by the sum of weights for all items in that component, and multiplying this number by 100. Component scores could range from 0-100, with a higher component score indicating greater disease burden. The Total score is calculated by summing the weights to all the positive responses in each component, dividing by the sum of weights for all items in the questionnaire, and multiplying this number by 100. SGRQ-C Total scores could range from 0-100, with a higher SGRQ-C Total score indicating greater disease burden. Participants were to assess their COPD symptoms, activity and impact at Baseline, Week 26, Week 52, and Week 104.
Time Frame: Baseline and Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Baseline and Week 26, Week 52 or Week 104 assessment for SGRQ-C score. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 130 | 112 | 106 | 131
Score on a Scale
  Change at Week 26 (n=130, 112, 106, 131) | -2.65 (1.15) | -2.28 (1.21) | -4.63 (1.23) | -1.60 (1.15)
  Change at Week 52 (n=62, 50, 45, 63) | -2.49 (1.58) | -2.22 (1.73) | -3.86 (1.80) | -4.40 (1.57)
  Change at Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

9. Secondary Outcome: Change From Baseline in Distance Walked in 6 Minutes (6-Minute Walk Test)
Description: The 6-minute walk test measures the distance participants can walk quickly on a flat, hard surface in 6 minutes. The 6-minute walk test was to be conducted at Baseline, Week 26, Week 52 and Week 104.
Time Frame: Baseline and Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants at selected sites who received at least one dose of study drug and had a Baseline and Week 26, Week 52 or Week 104 assessment for 6-minute walk test. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 84 | 77 | 68 | 87
Meters
  Change at Week 26 (n=84, 77, 68, 87) | 18.87 (6.55) | -1.04 (6.79) | 2.06 (7.19) | 7.41 (6.45)
  Change at Week 52 (n=32, 25, 25, 30) | 19.79 (11.50) | -33.58 (12.74) | 0.93 (12.84) | -15.37 (11.77)
  Change at Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

10. Secondary Outcome: Change From Baseline in Pre-bronchodilator FEV1
Description: FEV1, as measured in liters by spirometry, is the amount of air expired in 1 second. Pre-bronchodilator FEV1 was to be assessed immediately before bronchodilator administration at Baseline, Week 26, Week 52 and Week 104.
Time Frame: Baseline and Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Baseline and Week 26, Week 52 or Week 104 assessment for pre-bronchodilator FEV1. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 124 | 104 | 103 | 126
Liters
  Change at Week 26 (n=124, 104, 103 126) | -0.035 (0.021) | -0.084 (0.022) | 0.008 (0.022) | -0.054 (0.021)
  Change at Week 52 (n=65, 47, 43, 67) | -0.049 (0.025) | -0.084 (0.028) | 0.019 (0.029) | -0.073 (0.025)
  Change at Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

11. Secondary Outcome: Change From Baseline in Forced Expiratory Flow During the Middle Half of the Forced Vital Capacity (FEF25%-75%) Test
Description: Mid-Breath Forced Expiratory Flow (FEF25%-75%), as measured in liters/minute by spirometry, is the rate at which participants breathe out air from 25 percent of their breath to 75 percent of their breath. FEF25%-75% was to be assessed at Baseline, Week 26, Week 52 and Week 104.
Time Frame: Baseline and Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Baseline and Week 26, Week 52 or Week 104 assessment for FEF25%-75%. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 124 | 105 | 102 | 127
Liters/minute
  Change at Week 26 (n=124, 105, 102, 127) | 0.000 (0.016) | -0.053 (0.017) | 0.028 (0.017) | -0.022 (0.016)
  Change at Week 52 (n=66, 47, 44, 65) | -0.008 (0.020) | -0.055 (0.022) | 0.031 (0.023) | -0.018 (0.020)
  Change at Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

12. Secondary Outcome: Change From Baseline in Post-bronchodilator Forced Vital Capacity (FVC)
Description: FVC, as measured in liters by spirometry, is the amount of air forcibly exhaled from the lungs after taking the deepest breath possible. Post-bronchodilator FVC was to be assessed 30 minutes after bronchodilator administration (4 puffs of albuterol/salbutamol or equivalent separated by 30-second intervals) at Baseline, Week 26, Week 52 and Week 104.
Time Frame: Baseline and Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Baseline and Week 26, Week 52 or Week 104 assessment for post-bronchodilator FVC. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 124 | 105 | 102 | 127
Liters
  Change at Week 26 (n=124, 105, 102, 127) | -0.020 (0.040) | -0.089 (0.042) | -0.009 (0.043) | -0.086 (0.039)
  Change at Week 52 (n=66, 47, 44, 65) | -0.106 (0.050) | -0.077 (0.057) | 0.039 (0.059) | -0.057 (0.050)
  Change at Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

13. Secondary Outcome: Change From Baseline in Functional Residual Capacity (FRC)
Description: FRC, as measured in liters by body plethysmography, is the volume of air present in the lungs at the end of passive expiration. FRC was to be assessed after post-bronchodilator spirometry tests were performed at Baseline, Week 26, Week 52 and Week 104.
Time Frame: Baseline and Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Baseline and Week 26, Week 52 or Week 104 assessment for FRC. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 65 | 55 | 50 | 59
Liters
  Change at Week 26 (n=65, 55, 50, 59) | 0.15 (0.11) | -0.11 (0.12) | -0.07 (0.12) | 0.07 (0.11)
  Change at Week 52 (n=24, 21, 18, 21) | 0.21 (0.13) | 0.12 (0.14) | 0.10 (0.15) | 0.13 (0.14)
  Change at Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

14. Secondary Outcome: Change From Baseline in Total Lung Capacity (TLC)
Description: TLC, as measured in liters by body plethysmography, is the most amount of air lungs can hold at the top of breathing in. TLC was to be assessed after post-bronchodilator spirometry tests were performed at Baseline, Week 26, Week 52 and Week 104.
Time Frame: Baseline and Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Baseline and Week 26, Week 52 or Week 104 assessment for TLC. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 65 | 55 | 50 | 59
Liters
  Change at Week 26 (n=65, 55, 50, 59) | 0.11 (0.11) | -0.14 (0.12) | -0.06 (0.12) | 0.03 (0.11)
  Change at Week 52 (n=24, 21, 18, 21) | 0.15 (0.13) | 0.01 (0.14) | 0.13 (0.15) | 0.11 (0.14)
  Change at Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

15. Secondary Outcome: Change From Baseline in Inspiratory Capacity (IC)
Description: IC, as measured in liters by body plethysmography, is the maximum amount of air inspired when taking a slow, full inspiration with no hesitation from a position of passive end-tidal expiration (i.e. FRC) to a position of maximal inspiration. IC was to be assessed after post-bronchodilator spirometry tests were performed at Baseline, Week 26, Week 52 and Week 104.
Time Frame: Baseline and Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Baseline and Week 26, Week 52 or Week 104 assessment for IC. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 66 | 55 | 50 | 60
Liters
  Change at Week 26 (n=66, 55, 50, 60) | -0.04 (0.05) | -0.05 (0.06) | 0.01 (0.06) | -0.05 (0.06)
  Change at Week 52 (n=24, 21, 18, 21) | -0.02 (0.08) | -0.12 (0.09) | 0.04 (0.09) | 0.02 (0.09)
  Change at Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

16. Secondary Outcome: Change From Baseline in Morning Peak Expiratory Flow (PEF)
Description: PEF, as measured in liters/minute with a peak flow meter, is the maximum speed of expiration. Participants were to perform at least 3 and up to 5 PEF measurements in the morning before taking study drug. PEF was to be assessed at Baseline, Week 26, Week 52 and Week 104.
Time Frame: Baseline and Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Baseline and Week 26, Week 52 or Week 104 assessment for PEF. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 119 | 97 | 95 | 122
Liters/minute
  Change at Week 26 (n=119, 97, 95, 122) | -14.7 (4.28) | -20.5 (4.50) | -11.6 (4.61) | -21.8 (4.26)
  Change at Week 52 (n=61, 48, 43, 63) | -23.7 (9.69) | -22.9 (10.88) | -0.48 (11.50) | -26.2 (9.54)
  Change at Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

17. Secondary Outcome: Change From Baseline in Body-Mass Index, Airflow Obstruction, Dyspnea, and Exercise Capacity (BODE) Index Score
Description: The BODE index is a composite score assessing COPD prognosis that consists of 4 variables that are individually scored: FEV1 percent predicted, 6-Minute Walk Test, Modified Medical Research Council (MMRC) dyspnea scale and body mass index (BMI). The FEV1 percent predicted was scored from ≥65% (0 points, less airway obstruction) to ≤35% (3 points, greater airway obstruction). The 6-Minute Walk Distance was scored from: ≥350 meters (0 points, good exercise capacity) to ≤149 meters (3 points, poor exercise capacity). The MMRC Dyspnea Scale was scored from: MMRC 0: Dyspneic on strenuous exercise (0 points) to MMRC 4: Cannot leave house; breathless on dressing/undressing (3 points). BMI was scored as: >21 (0 points) and ≤21 (1 point). Variable scores were summed to produce a BODE index score. BODE index scores could range from 0 to 10, with a higher score correlating with an increased risk of COPD mortality. BODE index scores were to be assessed at Baseline, Week 26, Week 52 and Week 104.
Time Frame: Baseline and Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants at selected sites who received at least one dose of study drug and had a Baseline and Week 26, Week 52 or Week 104 assessment for BODE index score. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 83 | 72 | 67 | 84
Score on a Scale
  Change at Week 26 (n=83, 72, 67, 84) | -0.35 (0.12) | 0.13 (0.13) | -0.21 (0.13) | 0.07 (0.12)
  Change at Week 52 (n=31, 21, 23, 27) | -0.10 (0.21) | -0.02 (0.25) | 0.09 (0.24) | 0.12 (0.22)
  Change at Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

18. Secondary Outcome: Change From Baseline in Modified Medical Research Council (MMRC) Dyspnea Score
Description: The MMRC dyspnea scale is used to assess participant breathlessness. The MMRC dyspnea scale consists of five grades that describe almost the entire range of respiratory disability from none (Grade 0=Not troubled with breathlessness except with strenuous exercise) to almost complete incapacity (Grade 4=Too breathless to leave the house or breathless when dressing or undressing). MMRC dyspnea scores were to be assessed at Baseline, Week 26, Week 52 and Week 104.
Time Frame: Baseline and Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Baseline and Week 26, Week 52 or Week 104 assessment for MMRC dyspnea score. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 83 | 75 | 68 | 86
Score on a Scale
  Change at Week 26 (n=83, 75, 68, 86) | -0.34 (0.08) | -0.02 (0.09) | -0.24 (0.09) | -0.07 (0.08)
  Change at Week 52 (n=33, 28, 25, 31) | -0.25 (0.15) | 0.05 (0.16) | -0.09 (0.17) | -0.07 (0.15)
  Change at Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

19. Secondary Outcome: Sputum Inflammatory Marker Levels: Interleukin 8 (IL-8)
Description: Induced sputum samples were to be collected from participants via the nebulized method prior to study drug administration at Week 26, Week 52 and Week 104. IL-8 levels were measured by enzyme-linked immunosorbent assay (ELISA) in the sputum supernatant. The reported Baseline LS means and SDs are pooled across all treatment groups. The rationale for the use of pooled Baseline LS mean and SD values is the assumption that the Baseline LS mean and SD values are similar across treatment groups. The reported post-Baseline SDs are pooled across all treatment groups. The rationale for the use of an ANOVA method using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline, Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants at selected sites who received at least one dose of study drug and had a Week 26, Week 52 or Week 104 assessment for sputum IL-8 level. The study was terminated during Period 2; no data were collected for this endpoint at Weeks 52 or 104.
Measure: Least Squares Mean (Standard Deviation); unit: pg/mL
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 38 | 36 | 48 | 42
pg/mL
  Baseline (n=38, 36, 48, 42) | 29.736 (0.552) | 29.736 (0.552) | 29.736 (0.552) | 29.736 (0.552)
  Week 26 (n=24, 22, 19, 21) | 35.392 (0.410) | 38.471 (0.410) | 31.693 (0.410) | 30.421 (0.410)
  Week 52 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.
  Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

20. Secondary Outcome: Sputum Inflammatory Marker Levels: Myeloperoxidase (MPO)
Description: Induced sputum samples were to be collected from participants via the nebulized method prior to study drug administration at Week 26, Week 52 and Week 104. MPO levels were measured by ELISA in the sputum supernatant. The reported Baseline LS means and SDs are pooled across all treatment groups. The rationale for the use of pooled Baseline LS mean and SD values is the assumption that the Baseline LS mean and SD values are similar across treatment groups. The reported post-Baseline SDs are pooled across all treatment groups. The rationale for the use of an ANOVA method using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline, Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants at selected sites who received at least one dose of study drug and had a Week 26, Week 52 or Week 104 assessment for sputum MPO level. The study was terminated during Period 2; no data were collected for this endpoint at Weeks 52 or 104.
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 37 | 36 | 45 | 41
ng/mL
  Baseline (n=37, 36, 45, 41) | 1.840 (1.120) | 1.840 (1.120) | 1.840 (1.120) | 1.840 (1.120)
  Week 26 (n=24, 22, 19, 20) | 3.243 (1.488) | 1.747 (1.488) | 0.932 (1.488) | 3.656 (1.488)
  Week 52 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.
  Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

21. Secondary Outcome: Sputum Inflammatory Marker Levels: Sputum Neutrophil Elastase
Description: Induced sputum samples were to be collected from participants via the nebulized method prior to study drug administration at Week 26, Week 52 and Week 104. Neutrophil elastase levels were measured in the sputum supernatant. The reported Baseline LS means and SDs are pooled across all treatment groups. The rationale for the use of pooled Baseline LS mean and SD values is the assumption that the Baseline LS mean and SD values are similar across treatment groups. The reported post-Baseline SDs are pooled across all treatment groups. The rationale for the use of an ANOVA method using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline, Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants at selected sites who received at least one dose of study drug and had a Week 26, Week 52 or Week 104 assessment for sputum neutrophil elastase level. The study was terminated during Period 2; no data were collected for this endpoint at Weeks 52 or 104.
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 36 | 34 | 43 | 37
ng/mL
  Baseline (n=36, 34, 43, 37) | 16.948 (0.700) | 16.948 (0.700) | 16.948 (0.700) | 16.948 (0.700)
  Week 26 (n=23, 17, 19, 19) | 16.785 (0.773) | 11.365 (0.773) | 19.106 (0.773) | 27.973 (0.773)
  Week 52 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.
  Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

22. Secondary Outcome: Sputum Inflammatory Marker Levels: Matrix Metallopeptidase-9 (MMP-9)
Description: Induced sputum samples were to be collected from participants via the nebulized method prior to study drug administration at Week 26, Week 52 and Week 104. MMP-9 levels were measured by ELISA in the sputum supernatant. The reported Baseline LS means and SDs are pooled across all treatment groups. The rationale for the use of pooled Baseline LS mean and SD values is the assumption that the Baseline LS mean and SD values are similar across treatment groups. The reported post-Baseline SDs are pooled across all treatment groups. The rationale for the use of an ANOVA method using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline, Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants at selected sites who received at least one dose of study drug and had a Week 26, Week 52 or Week 104 assessment for induced sputum MMP-9 level. The study was terminated during Period 2; no data were collected for this endpoint at Weeks 52 or 104.
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 39 | 35 | 46 | 41
ng/mL
  Baseline (n=39, 35, 46, 41) | 720.45 (0.773) | 720.45 (0.773) | 720.45 (0.773) | 720.45 (0.773)
  Week 26 (n=24, 22, 19, 21) | 878.02 (0.709) | 711.90 (0.709) | 392.81 (0.709) | 1480.1 (0.709)
  Week 52 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.
  Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

23. Secondary Outcome: Plasma Inflammatory Biomarker Levels: High-sensitivity C-reactive Protein (Hs-CRP)
Description: Blood samples were to be collected prior to study drug administration to determine participant plasma hs-CRP levels at Week 26, Week 52 and Week 104. The reported Baseline LS means and SDs are pooled across all treatment groups. The rationale for the use of pooled Baseline LS mean and SD values is the assumption that the Baseline LS mean and SD values are similar across treatment groups. The reported post-Baseline SDs are pooled across all treatment groups. The rationale for the use of an ANOVA method using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline, Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Week 26, Week 52 or Week 104 assessment for plasma hs-CRP level. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Deviation); unit: mg/dL
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 148 | 152 | 149 | 150
mg/dL
  Baseline (n=148, 152, 149, 150) | 2.766 (0.498) | 2.766 (0.498) | 2.766 (0.498) | 2.766 (0.498)
  Week 26 (n=121, 104, 100, 126) | 2.832 (0.443) | 3.728 (0.443) | 4.410 (0.443) | 2.889 (0.443)
  Week 52 (n=67, 49, 43, 68) | 3.360 (0.432) | 3.871 (0.432) | 4.566 (0.432) | 2.657 (0.432)
  Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

24. Secondary Outcome: Plasma Inflammatory Biomarker Levels: Fibrinogen
Description: Blood samples were to be collected prior to study drug administration to determine participant plasma fibrinogen levels at Week 26, Week 52 and Week 104. The reported Baseline LS means and SDs are pooled across all treatment groups. The rationale for the use of pooled Baseline LS mean and SD values is the assumption that the Baseline LS mean and SD values are similar across treatment groups. The reported post-Baseline SDs are pooled across all treatment groups. The rationale for the use of an ANOVA method using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline, Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Week 26, Week 52 or Week 104 assessment for plasma fibrinogen level. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Deviation); unit: mg/dL
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 140 | 138 | 138 | 143
mg/dL
  Baseline (n=140, 138, 138, 143) | 3.731 (0.108) | 3.731 (0.108) | 3.731 (0.108) | 3.731 (0.108)
  Week 26 (n=111, 104, 91, 121) | 3.835 (0.119) | 4.027 (0.119) | 4.068 (0.119) | 3.788 (0.119)
  Week 52 (n=52, 40, 38, 58) | 4.163 (0.108) | 4.031 (0.108) | 4.308 (0.108) | 3.788 (0.108)
  Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

25. Secondary Outcome: Plasma Inflammatory Biomarker Levels: Myeloperoxidase (MPO)
Description: Blood samples were to be collected prior to study drug administration to determine participant plasma MPO levels at Week 26, Week 52 and Week 104. The reported Baseline LS means and SDs are pooled across all treatment groups. The rationale for the use of pooled Baseline LS mean and SD values is the assumption that the Baseline LS mean and SD values are similar across treatment groups. The reported post-Baseline SDs are pooled across all treatment groups. The rationale for the use of an ANOVA method using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline, Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Week 26, Week 52 or Week 104 assessment for MPO level. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 146 | 145 | 147 | 148
ng/mL
  Baseline (n=146, 145, 147, 148) | 169.15 (0.386) | 169.15 (0.386) | 169.15 (0.386) | 169.15 (0.386)
  Week 26 (n=119, 104, 97, 124) | 188.70 (0.439) | 175.80 (0.439) | 173.16 (0.439) | 227.72 (0.439)
  Week 52 (n=47, 36, 35, 46) | 234.42 (0.451) | 196.67 (0.451) | 246.04 (0.451) | 254.20 (0.451)
  Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

26. Secondary Outcome: Plasma Inflammatory Biomarker Levels: Matrix Metallopeptidase-9 (MMP-9)
Description: Blood samples were to be collected prior to study drug administration to determine participant plasma MMP-9 levels at Week 26, Week 52 and Week 104. The reported Baseline LS means and SDs are pooled across all treatment groups. The rationale for the use of pooled Baseline LS mean and SD values is the assumption that the Baseline LS mean and SD values are similar across treatment groups. The reported post-Baseline SDs are pooled across all treatment groups. The rationale for the use of an ANOVA method using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline, Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Week 26, Week 52 or Week 104 assessment for MMP-9 level. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 146 | 145 | 147 | 148
ng/mL
  Baseline (n=146, 145, 147, 148) | 294.80 (0.254) | 294.80 (0.254) | 294.80 (0.254) | 294.80 (0.254)
  Week 26 (n=119, 104, 97, 124) | 247.63 (0.272) | 216.40 (0.272) | 217.79 (0.272) | 319.80 (0.272)
  Week 52 (n=48, 36, 35, 47) | 258.82 (0.272) | 220.90 (0.272) | 244.67 (0.272) | 342.46 (0.272)
  Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

27. Secondary Outcome: Plasma Inflammatory Biomarker Levels: Plasma Neutrophil Elastase
Description: Blood samples were to be collected prior to study drug administration to determine participant plasma neutrophil elastase levels at Week 26, Week 52 and Week 104. The reported Baseline LS means and SDs are pooled across all treatment groups. The rationale for the use of pooled Baseline LS mean and SD values is the assumption that the Baseline LS mean and SD values are similar across treatment groups. The reported post-Baseline SDs are pooled across all treatment groups. The rationale for the use of an ANOVA method using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline, Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Week 26, Week 52 or Week 104 assessment for plasma neutrophil elastase level. The study was terminated during Period 2; no data were collected for the endpoint at Week 104.
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 123 | 117 | 122 | 121
ng/mL
  Baseline (n=123, 117, 122, 121) | 67.969 (0.323) | 67.969 (0.323) | 67.969 (0.323) | 67.969 (0.323)
  Week 26 (n=118, 104, 93, 121) | 63.592 (0.341) | 63.680 (0.341) | 65.413 (0.341) | 67.697 (0.341)
  Week 52 (n=51, 41, 33, 52) | 60.965 (0.280) | 54.267 (0.280) | 64.296 (0.280) | 57.804 (0.280)
  Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

28. Secondary Outcome: Plasma Inflammatory Biomarker Levels: Epithelial Cell-Derived Neutrophil Activating Peptide 78 (ENA-78)
Description: Blood samples were to be collected prior to study drug administration to determine participant plasma ENA-78 levels at Week 26, Week 52 and Week 104. The reported Baseline LS means and SDs are pooled across all treatment groups. The rationale for the use of pooled Baseline LS mean and SD values is the assumption that the Baseline LS mean and SD values are similar across treatment groups. The reported post-Baseline SDs are pooled across all treatment groups. The rationale for the use of an ANOVA method using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline, Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants who received at least one dose of study drug and had a Week 26, Week 52 or Week 104 assessment for ENA-78 level. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Deviation); unit: pg/mL
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 125 | 118 | 122 | 126
pg/mL
  Baseline (n=125, 118, 122, 126) | 436.31 (0.430) | 436.31 (0.430) | 436.31 (0.430) | 436.31 (0.430)
  Week 26 (n=119, 105, 92, 121) | 508.31 (0.451) | 543.60 (0.451) | 607.37 (0.451) | 473.10 (0.451)
  Week 52 (n=42, 32, 33, 42) | 509.93 (0.409) | 603.44 (0.409) | 698.93 (0.409) | 417.90 (0.409)
  Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

29. Secondary Outcome: Change From Baseline in Pre- and Post-6-Minute-Walk-Test Borg Scale Score
Description: The 6-minute walk test measured the distance participants could walk quickly on a flat, hard surface in 6 minutes. The Borg scale is a method use to rate perceived exertion (0=Nothing at all [no exertion] to 10=Maximal [exertion]). Borg scale scores were to be assessed pre- and post-walk-test at Baseline, Week 26, Week 52 and Week 104. A higher score indicates greater perceived exertion.
Time Frame: Baseline and Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants at selected sites who received at least one dose of study drug and had a Baseline and Week 26, Week 52 or Week 104 assessment for pre- and post-6-minute-walk-test Borg scale score. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 84 | 77 | 68 | 87
Score on a Scale
  Pre-walk Change at Week 26 (n=84, 77, 68, 87) | -0.27 (0.12) | 0.07 (0.12) | -0.13 (0.13) | 0.17 (0.12)
  Pre-walk Change at Week 52 (n=32, 25, 25, 30) | -0.18 (0.19) | 0.22 (0.21) | 0.08 (0.21) | 0.21 (0.20)
  Post-walk Change at Week 26 (n=84, 77, 68, 87) | -0.52 (0.14) | -0.03 (0.15) | 0.10 (0.16) | 0.11 (0.14)
  Post-walk Change at Week 52 (n=32, 25, 25, 30) | -0.26 (0.26) | 0.52 (0.29) | -0.16 (0.30) | 0.26 (0.27)
  Pre-walk Change at Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.
  Post-walk Change at Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

30. Secondary Outcome: Change From Baseline in Percent of Arterial Oxygen Saturation Measured by Pulse Oximetry Before and After the 6-Minute Walk Test
Description: The 6-minute walk test measured the distance participants could walk quickly on a flat, hard surface in 6 minutes. Percent (%) of arterial oxygen saturation, as measured by pulse oximetry, was to be assessed before and after the 6-minute walk test at Baseline, Week 26, Week 52 and Week 104.
Time Frame: Baseline and Week 26, Week 52, Week 104
Population: The FAS population consisted of all participants at selected sites who received at least one dose of study drug and had a Baseline and Week 26, Week 52 or Week 104 assessment for pre- and post-6-minute-walk-test arterial oxygen saturation. The study was terminated during Period 2; no data were collected for this endpoint at Week 104.
Measure: Least Squares Mean (Standard Error); unit: Percent Oxygen Saturation
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 84 | 77 | 68 | 87
Percent Oxygen Saturation
  Pre-walk Change at Week 26 (n=84, 77, 68, 87) | 0.12 (0.21) | -0.70 (0.22) | -0.07 (0.23) | -0.02 (0.21)
  Pre-walk Change at Week 52 (n=32, 25, 25, 30) | 0.19 (0.32) | -0.08 (0.36) | -0.22 (0.36) | -0.00 (0.33)
  Post-walk Change at Week 26 (n=84, 77, 68, 87) | 0.26 (0.32) | -0.42 (0.33) | 0.28 (0.35) | 0.75 (0.32)
  Post-walk Change at Week 52 (n=32, 25, 25, 30) | 0.39 (0.45) | -0.33 (0.49) | 0.63 (0.50) | 0.19 (0.46)
  Pre-walk Change at Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.
  Post-walk Change at Week 104 (n=0, 0, 0, 0) | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected. | NA (NA) — Study terminated; data not collected.

31. Secondary Outcome: Percentage of Participants Who Experienced an AE Related to Respiratory Infection
Description: The percentage of participants who experienced an AE related to a respiratory infection or infestation, was to be calculated for the first 26 weeks, the first 52 weeks and the first 104 weeks of treatment.
Time Frame: Up to 26 , 52 and 104 weeks
Population: The ASaT population consisted of all participants who received at least one dose of study drug. The study was terminated during Period 2; no data were analyzed for this endpoint for up to 104 weeks.
Measure: Number; unit: Percentage of Participants
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 152 | 156 | 152 | 154
Percentage of Participants
  Up to Week 26 (n=152, 165, 152, 154) | 30.3 | 30.1 | 22.4 | 24.0
  Up to Week 52 (n=75, 63, 55, 82) | 41.3 | 41.3 | 38.2 | 28.0
  Up to Week 104 (n=0, 0, 0, 0) | NA — Study terminated; data not analyzed. | NA — Study terminated; data not analyzed. | NA — Study terminated; data not analyzed. | NA — Study terminated; data not analyzed.

32. Secondary Outcome: Percentage of Participants Who Experienced an AE Related to Any Type of Infection
Description: The percentage of participants who experienced an AE related to any type of infection or infestation, was to be calculated for the first 26 weeks, the first 52 weeks and the first 104 weeks of treatment.
Time Frame: Up to 26 , 52 and 104 weeks
Population: as for outcome 31
Measure: Number; unit: Percentage of Participants
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Number analyzed (Participants) | 152 | 156 | 152 | 154
Percentage of Participants
  Up to Week 26 (n=152, 156, 152, 154) | 34.2 | 37.2 | 27.0 | 31.8
  Up to Week 52 (n=75, 63, 55, 82) | 48.0 | 46.0 | 45.5 | 35.4
  Up to Week 104 (n=0, 0, 0, 0) | NA — Study terminated; data not analyzed. | NA — Study terminated; data not analyzed. | NA — Study terminated; data not analyzed. | NA — Study terminated; data not analyzed.

ADVERSE EVENTS:
Time Frame: Up to one week after last dose of study drug (up to 105 weeks)
Description: The ASaT population consisted of all participants who received at least one dose of study drug.
Arm/Group | Navarixin 10 mg | Navarixin 30 mg | Navarixin 50 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 26/152 | 23/156 | 20/152 | 21/154
Other Adverse Events (participants affected / at risk) | 65/152 | 75/156 | 74/152 | 46/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Navarixin 10 mg (N=152) | Navarixin 30 mg (N=156) | Navarixin 50 mg (N=152) | Placebo (N=154)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Megacolon (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4) | 2 (2) | 5 (5)
Scrotal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriogram coronary (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cancer Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 5 (6) | 6 (6) | 4 (10)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial bypass operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Navarixin 10 mg (N=152) | Navarixin 30 mg (N=156) | Navarixin 50 mg (N=152) | Placebo (N=154)
Influenza (Infections and infestations) | 9 (11) | 3 (3) | 4 (4) | 4 (6)
Nasopharyngitis (Infections and infestations) | 23 (38) | 28 (42) | 22 (34) | 22 (29)
Rhinitis (Infections and infestations) | 8 (8) | 6 (7) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 8 (11)
Overdose (Injury, poisoning and procedural complications) | 4 (5) | 4 (4) | 8 (9) | 4 (4)
Neutrophil count decreased (Investigations) | 6 (6) | 22 (22) | 32 (32) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 6 (7) | 8 (9) | 1 (1)
Headache (Nervous system disorders) | 14 (27) | 20 (29) | 14 (21) | 15 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including, without limitation, slides and texts of oral or other public presentations and texts of any transmission through any electronic media, e.g., any computer access system such as the Internet, World Wide Web, etc.) that report any results of the study.